CLINICAL TRIAL: NCT00114712
Title: The Ribavirin Pregnancy Registry
Acronym: RPR
Status: Terminated | Type: Observational
Why Stopped: Per the Division of Project Management, Office of Regulatory Operations, Office of Generic Drugs, FDA there is no regulatory requirement to continue this Registry.
Sponsor: Syneos Health (Other)
Collaborators: Aurobindo Pharma Ltd (Industry); Sandoz (Industry); Merck Sharp & Dohme LLC (Industry); Teva Pharmaceuticals USA (Industry); Zydus Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RPR-1
Record Dates: First submitted 2005-06-16; First posted 2005-06-17 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-03

CONDITIONS: Birth Defects; Pregnancy Complications; Hepatitis C
Keywords: Birth Defects; Pregnancy; Ribavirin; Hepatitis C
MeSH Terms: conditions — Congenital Abnormalities; Pregnancy Complications; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ribavirin should be avoided during pregnancy and during the 6 months before pregnancy in both the female and the male sexual partner. If a pregnancy occurs and is reported to the Ribavirin Pregnancy Registry, the Registry will follow the pregnant woman throughout pregnancy. The Registry will also follow the infant until 1 year of age. The goal of the Registry is to learn more about the effects of ribavirin on pregnancy and the risk for birth defects. Pregnant women exposed to ribavirin, either by taking ribavirin (during pregnancy or 6 months before pregnancy) or through a male sexual partner (who took ribavirin during the female partner's pregnancy or during the 6 months before pregnancy), are encouraged to contact the Registry.

DETAILED DESCRIPTION:
Ribavirin, a nucleoside analog with antiviral activity, is used in combination with interferons or pegylated interferons for the treatment of chronic hepatitis C (HCV). Extensive clinical studies have demonstrated that combination therapy with ribavirin and interferons or pegylated interferons are efficacious treatments for HCV. However, ribavirin has been assigned a FDA Pregnancy Category X classification, indicating that it should not be used in women who are pregnant or in men whose partners may become pregnant. Because the incidence of HCV is highest in the group with the highest reproductive potential, the 25 - 45 year age group, (CDC, 2001) it is likely that inadvertent pregnancy exposures will occur and should be monitored. The primary objectives of this Registry are:

* To evaluate the association between ribavirin and birth defects occurring in offspring of female patients exposed to ribavirin during pregnancy or within six months after therapy has stopped.
* To evaluate the association between ribavirin and birth defects occurring in offspring of females exposed to ribavirin during pregnancy or within six months after therapy has stopped, through their male sexual partners taking ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy occurring to one of the following groups while the patient or sexual partner was on ribavirin and/or within six months after therapy stopped:

  * Female patients who become pregnant on ribavirin therapy, or
  * Female patients who start ribavirin therapy while pregnant, or
  * Female patients who become pregnant post-ribavirin therapy (defined as the six month time period after therapy has stopped) or
  * Females who become pregnant while their male sexual partner is on ribavirin therapy or
  * Females who are pregnant when their male sexual partner starts ribavirin therapy, or
  * Females who become pregnant while their male sexual partner is in the post-ribavirin therapy period (defined as the six month time period after therapy has stopped).
* Timing of the prenatal exposure to ribavirin, no broader than within six months prior to pregnancy or trimester during which the exposure took place.
* Sufficient information to determine whether the pregnancy is prospectively registered (i.e., whether the outcome of pregnancy was known at the time of the report).
* Date the pregnancy exposure report is registered.
* Source of the report (health care professional, pregnant patient, or male sexual partner).
* Report contact information to allow for follow-up.

Exclusion Criteria:

* Females who were not exposed to Ribavirin during the designated time (described above)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Analysis - US
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2004-01; Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
To evaluate association between ribavirin and birth defects | At birth outcome, infant follow-up at 6 and 12 months
  To evaluate the association between ribavirin and birth defects occurring in offspring of female patients exposed to ribavirin during pregnancy or within six months after therapy has stopped.
  To evaluate the association between ribavirin and birth defects occurring in offspring of females exposed to ribavirin during pregnancy or within six months after therapy has stopped, through their male sexual partners taking ribavirin.

SECONDARY OUTCOMES:
Estimate risk of birth defects in exposed pregnancies | At birth outcome, infant follow-up at 6 and 12 months
  Attempt to estimate the risk of birth defects occurring in offspring of female patients exposed to ribavirin during pregnancy or within six months after therapy has stopped, and detect any increase in the prevalence or pattern of birth defects among these pregnancies.
  Attempt to estimate the risk of birth defects occurring in offspring of females exposed to ribavirin during pregnancy or within six months after therapy has stopped, through their male sexual partners taking ribavirin, to detect any increase in the prevalence or pattern of birth defects among these pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sinclair, PhD, Principal Investigator — Syneos Health
Locations (1):
- INC Research, LLC, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A condensed version of the annual interim report is available to healthcare providers upon request.

REFERENCES:
- [Derived] Sinclair SM, Jones JK, Miller RK, Greene MF, Kwo PY, Maddrey WC. The Ribavirin Pregnancy Registry: An Interim Analysis of Potential Teratogenicity at the Mid-Point of Enrollment. Drug Saf. 2017 Dec;40(12):1205-1218. doi: 10.1007/s40264-017-0566-6. PMID 28689333